CLINICAL TRIAL: NCT04465175
Title: Single Versus Double Dose Magnisum Sulphate in the Treatment of Moderate to Severe Asthma in Children in the Emergency Department
Brief Title: Double Dose Magnesium Sulphate in Moderate-severe Asthma in Paediatrics
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Noora Nasser Al-Alawi, Emergency resident -Oman medical specialty board, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mag4As
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Asthma in Children
Keywords: asthma , Magnesium sulphate
MeSH Terms: conditions — Asthma | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second dose magnesium sulphate (Active Comparator): Second dose magnesium sulphate 50 mg/kg infused over one hour
  Interventions: Drug: Magnesium Sulfate
- Placebo (Placebo Comparator): Normal saline (2.5 ml/kg) infused over one hour
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Sulfate — Second dose magnesium sulphate infusion over one hour
  Other Names: MgSO4
  Arms: Second dose magnesium sulphate
Drug: Placebo — Normal saline (2.5 ml/kg) infusion over one hour
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Introduction : . In Oman the prevalence of asthma was estimated to be 7.3% of adults and 12.7% of children . Magnesium sulphate is the second line treatment, many studies had shown that it has beneficial effect in treating acute asthma in children ; it reduces the hospital stay and the rate of admission as well as the ventilation rate .

Aim : To compare single dose Magnesium sulphate that is typically given in the emergency department verses two doses of magnesium sulphate in treating acute moderate-severe asthma exacerbation in paediatric age group Research hypothesis : Children who are treated with two doses MgSO4 are more likely to have improvement in their PRAM score and are less likely to be admitted to the ward, HD or ICU Primary outcome : Improvement in PRAM (Paediatric respiratory assessment measure) score of acute asthma exacerbation Secondary outcome : Reduce admission rate to general ward, PICU and HD . Demonstrate the safety profile of double dose of magnesium sulphate.

Study Design : prospective blinded randomized trial

Study population : children age 3-13 years who presented to Royal hospital paediatric emergency with moderate-severe acute asthma

Intervention : two doses magnesium sulphate

Comparison : Placebo

Outcome : Improvement in PRAM score

DETAILED DESCRIPTION:
Research questions :

In children 3 to 13 years of age presenting to the pediatric emergency room with moderate to severe asthma exacerbation, does double dose Magnesium sulfate improve asthma severity (PRAM) score and reduce admission rate more than single dose?

Study design :

Prospective double-blinded randomized clinical trial in paediatric (from age 3-13 years) who presents to the emergency department (ED) at Sultan Royal hospital with moderate to severe Acute asthma (PRAM score >=5) , Consent will be obtained from the parents. Eligible subjects will be enrolled Control Group Will receive second dose magnesium sulphate (50 mg/kg over 1 hour = 2.5mllkg) Intervention Group Will receive Normal saline (2.5ml/kg over 1 hour )

Sample size:

90 patient will be needed ( 45 on each arm) to have 60% power to detect a difference on PRAM score between the groups at the 5% alpha (significance) level.

Study steps:

1. Initial nursing triage for all acute asthma exacerbation , initial PRAM score will be recorded
2. Initial standard management as per protocol , which includes :

   1. Oxygen if indicated
   2. Back to back salbutamol (2.5-5 mg) and ipratropium (0.25-0.5 mg )nebulization OR salbutamol MDI 5 puffs (wt 10 Kg) -
   3. Systemic corticosteroid : children with PRAM 5-8 give oral dexamethasone 0.3 mg/kg , those with PRAM score 9-12 give hydrocortisone 4 mg/kg IV
3. Child will reassessed after the initial measures , PRAM score will be recorded in the patient sheet
4. All children with persistent PRAM score of ≥ 5 will receive the first dose of magnesium sulphate ( 50 mg/kg over 20 minutes
5. After 30 minutes of the first dose Magnesium sulphate PRAM score will be recorded, during this period child will be given 20ml/hr normal saline
6. Children with persistent PRAM score ≥ 5 will be included in the study provided they met the inclusion and exclusion criteria (as mentioned below ) ,consent will be obtained from parents
7. If the child met the inclusion and exclusion criteria , the treating physician will pick one envelope from the research box , each envelope will have serial or sequencing number for the medications (saline or MgSO4 )
8. The pharmacist will prepare a 100 ml bags that contains either saline or 2 grams magnesium sulphate in 100ml. The content will be concealed from the treating physician by the pharmacist.
9. Child be will given 2.5 ml/kg from any bag chosen (based on the sequencing) . The total amount will be infused over one hour.
10. PRAM score post intervention will be recorded . Disposition will be based on physician assessment and improvement in PRAM score
11. Safety Assessments : All adverse events will be documented on an side effect section on patient's sheet case . Serious adverse events should be immediately reported to the primary investigator. Any serious, adverse event will be reported immediately to the Institutional Review Board.

Reported side effects for magnesium sulphte : nausea ,facial warmth , flushing , pain and numbness at infusion site , dry mouth and malaise . Rare side effect : hypotension

Beneficiaries of the research :

* To the child :

  * Improvement in his/her symptoms
  * Reduce PICU admission and intubation
  * Reduce the abstinences from school and improve the quality of life
* To the health system:

  * Availability of PICU and HDU beds for more sick patients
  * Reducing the cost of asthmatic patient care

ELIGIBILITY:
Inclusion Criteria:

* Physican diagnosed of asthma
* Age 3-13 years
* Children presenting with acute moderate- severe asthma (PRAM score ≥ 5)
* Failed to respond to initial treatment of acute asthma
* Not known to have allergy from MgSO4

Exclusion Criteria:

* Mild exacerbation of asthma (initial PRAM score ≤4)
* Other comorbid present : Significant heart disease , arrhythmias , chronic kidney disease , cystic fibrosis , operated trachea-esophageal fistula , known or operated for vascular ring , trisomy 21

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in PRAM (Paediatric respiratory assessment measure) score of acute asthma | at 60 minutes of intervention
  Improvement in PRAM (Paediatric respiratory assessment measure) score of acute asthma exacerbation

SECONDARY OUTCOMES:
Reduce admission rate to general ward, paediatric intensive care unit and high dependency unit | during first 24 hours
  Reduce admission rate to general ward, paediatric intensive care unit and high dependency unit
Demonstrate the safety profile of double dose of magnesium sulphate. | during first 24 hours
  Any side effects from giving second doses Magnesium sulphate

CONTACTS AND LOCATIONS:
Overall Officials: Noora Al-Alawi, Resident, Principal Investigator — Oman Medical Specialty Board

IPD SHARING:
Plan to Share IPD: No